CLINICAL TRIAL: NCT05485896
Title: A Prospective Single-arm Clinical Study of Pembrolizumab Combined With Lenvatinib Neoadjuvant Therapy in Patients With Advanced Renal Cell Carcinoma
Brief Title: Neoadjuvant Therapy of Pembrolizumab Plus Lenvatinib in Advanced RCC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tianjin Medical University Second Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PELUR
Record Dates: First submitted 2022-07-25; First posted 2022-08-03 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Renal Cell Carcinoma
Keywords: Pembrolizumab; Lenvatinib; Advanced Renal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — pembrolizumab; lenvatinib

STUDY DESIGN:
Intervention Model Description: Single Group Assignment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Advanced RCC (Locally advanced, regional LN invaded, or M1-NED) (Experimental): Patients will receive treatment with Pembrolizumab in combination with Lenvatinib every 3 weeks for 3 cycles in the preoperation. In addition, 17 cycles' Pembrolizumab were needed for patients with high risk of recurrence (tumor stage 2 with nuclear grade IV or sarcomatoid differentiation, tumor stage 3 or higher, regional lymph-node metastasis, or stage M1 with no evidence of disease residual).
  Interventions: Drug: Pembrolizumab plus Lenvatinib

INTERVENTIONS:
Drug: Pembrolizumab plus Lenvatinib — Patients will receive treatment with Pembrolizumab in combination with Lenvatinib every 3 weeks for 3 cycles in the preoperation. Additional 17 cycles of Pembrolizumab were needed for patients with high risk of recurrence (tumor stage 2 with nuclear grade IV or sarcomatoid differentiation, tumor stage 3 or higher, regional lymph-node metastasis, or stage M1 with no evidence of disease residual).

SUMMARY:
This is a phase II study to determine the efficacy and safety of Pembrolizumab when given in combination with Lenvatinib as treatment for patients with the advanced kidney cancer. Further evaluate whether the treatment plan is beneficial to the patient's surgery.

DETAILED DESCRIPTION:
This is a phase II study to determine the efficacy and safety of Pembrolizumab when given in combination with Lenvatinib as treatment for patients with the advanced kidney cancer . Further evaluate whether the treatment is beneficial to operation. Patients will receive treatment with Pembrolizumab in combination with Lenvatinib every 3 weeks for 3 cycles in the preoperation. Additional 17 cycles of Pembrolizumab were needed for patients with high risk of recurrence (tumor stage 2 with nuclear grade IV or sarcomatoid differentiation, tumor stage 3 or higher, regional lymph-node metastasis, or stage M1 with no evidence of disease residual).

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to provide written informed consent;
2. Age ≥ 18 years and age ≤75years;
3. Patients with pathologically and radiographically confirmed clear cell renal cell carcinoma with clinical staging: cTanyN1Many, cTanyNanyM1, cT3-4NanyMany, and all visible lesions could be excised or ablation treated;
4. Enhanced imaging evaluation can be performed;
5. There are no suspected brain metastases;
6. The presence of measurable lesions was assessed according to RECISTv1.1 criteria;
7. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-1;
8. Organ function level must meet the following requirements:

   Hematological indexes: neutrophil count >= 1.5x10^9/L, platelet count >= 100x10^9/L, hemoglobin >= 9.0 g/dl (can be maintained by blood transfusion); Liver function: total bilirubin <=1.5 ULN, alanine aminotransferase and aspartate aminotransferase <=1.5 ULN;
9. Women were required to use an effective contraceptive method for three months after the end of the study, and men were required to consent to use an effective contraceptive method with their spouse during and for three months after the end of the study;
10. The subjects volunteered to join the study, signed informed consent, and had good compliance with follow-up.

Exclusion Criteria:

1. Prior treatment with radiation, chemotherapy, long-term or high-dose hormone therapy, or immune checkpoint inhibitors;
2. Previous or concurrent other malignancy;
3. Previous PD-L1 or PD-L1 treatment, or allergy to PD-L1;
4. History of primary immunodeficiency;
5. Active, known or suspected autoimmune diseases;
6. Known history of allogeneic organ transplantation and allogeneic hematopoietic stem cell transplantation;
7. Pregnant or lactating female patients;
8. Untreated acute or chronic active hepatitis B or hepatitis C infection. Under the condition of monitoring the virus copy number of patients receiving antiviral treatment, doctors can judge whether they are in line with the patients' individual conditions;
9. Have a clear history of active tuberculosis;
10. Participating in other clinical researchers;
11. Men with reproductive capacity or women who are likely to become pregnant do not take reliable contraceptive measures;
12. Uncontrolled concurrent diseases, including but not limited to:

HIV infected (HIV antibody positive); Severe infection in active stage or poorly controlled; Evidence of serious or uncontrollable systemic diseases (such as severe mental, neurological, epilepsy or dementia, unstable or uncompensated respiratory, cardiovascular, liver or kidney diseases, uncontrolled hypertension [i.e. hypertension greater than or equal to CTCAE grade 2 after drug treatment]); Patients with active bleeding or new thrombotic disease.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-09-02 (Actual)

PRIMARY OUTCOMES:
Tumor responses | Through treatment completion (before surgery), an average of 3 cycles (each cycle is 21 days).
  All patients had imaging (enhanced CT, enhanced MRI or both ) before and after treatment to evaluate radiographic response within the primary tumor and venous tumor thrombus by using RECIST (Response Evaluation Criteria in Solid Tumors)
Adverse events | Through treatment completion (before surgery), an average of 3 cycles (each cycle is 21 days).
  Adverse events were monitored throughout treatment until 30 days after surgery and were evaluated according to Common Terminology Criteria for Adverse Events (version 5.0).

SECONDARY OUTCOMES:
Tumor viability assessment | Through treatment completion (before surgery), an average of 3 cycles (each cycle is 21 days).
  Densitometric measurement of tumor viability using a modification of the Choi criteria was performed to evaluate the effect. Briefly, using axial source computed tomography images (1.5 mm thickness) a three-dimensional image of the kidney was reconstructed with an imaging workstation (Terra Recon, San Mateo, CA).
Progression free survival | Every 12 weeks until 12 months after surgery
  Progression free survival was assessed by imaging (enhanced CT, enhanced MRI or both ) after surgery every 12 weeks until 12 months.

OTHER OUTCOMES:
Rate of responser with predictive biomarker positive | Through treatment completion (before surgery), an average of 3 cycles (each cycle is 21 days).
  Bulk RNA-seq and/or single cell RNA-seq were performed in part of tissues before and after neoadjuvant treatment to seek biomarkers predicting Response.

CONTACTS AND LOCATIONS:
Overall Officials: Changyi Quan, MD, Principal Investigator — Tianjin Medical University Second Hospital
Locations (1):
- Changyi Quan, Tianjin, Tianjin Municipality, China

REFERENCES:
- [Background] Motzer R, Alekseev B, Rha SY, Porta C, Eto M, Powles T, Grunwald V, Hutson TE, Kopyltsov E, Mendez-Vidal MJ, Kozlov V, Alyasova A, Hong SH, Kapoor A, Alonso Gordoa T, Merchan JR, Winquist E, Maroto P, Goh JC, Kim M, Gurney H, Patel V, Peer A, Procopio G, Takagi T, Melichar B, Rolland F, De Giorgi U, Wong S, Bedke J, Schmidinger M, Dutcus CE, Smith AD, Dutta L, Mody K, Perini RF, Xing D, Choueiri TK; CLEAR Trial Investigators. Lenvatinib plus Pembrolizumab or Everolimus for Advanced Renal Cell Carcinoma. N Engl J Med. 2021 Apr 8;384(14):1289-1300. doi: 10.1056/NEJMoa2035716. Epub 2021 Feb 13. PMID 33616314
- [Background] Choueiri TK, Tomczak P, Park SH, Venugopal B, Ferguson T, Chang YH, Hajek J, Symeonides SN, Lee JL, Sarwar N, Thiery-Vuillemin A, Gross-Goupil M, Mahave M, Haas NB, Sawrycki P, Gurney H, Chevreau C, Melichar B, Kopyltsov E, Alva A, Burke JM, Doshi G, Topart D, Oudard S, Hammers H, Kitamura H, Bedke J, Perini RF, Zhang P, Imai K, Willemann-Rogerio J, Quinn DI, Powles T; KEYNOTE-564 Investigators. Adjuvant Pembrolizumab after Nephrectomy in Renal-Cell Carcinoma. N Engl J Med. 2021 Aug 19;385(8):683-694. doi: 10.1056/NEJMoa2106391. PMID 34407342